CLINICAL TRIAL: NCT02427789
Title: Therapeutic Effectiveness of Exercise Associated to the Pharmacotherapy in Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCLim27/FAPESP2012/20002-5
Record Dates: First submitted 2014-01-24; First posted 2015-04-28 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2013-01

CONDITIONS: Major Depressive Disorder
Keywords: Physical exercise; Biomarkers; Neuroprotection; ergospirometry; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): In this group patients will not have physical exercises
- Physical Exercise (Active Comparator): In this group patients will make physical exercise
  Interventions: Other: Physical Exercise

INTERVENTIONS:
Other: Physical Exercise — physical exercise
  Arms: Physical Exercise

SUMMARY:
Depression is a disorder that causes major harm to physical health and social life. It induces isolation, reduced physical and work capacity and increasing the risk of death. In contrast, exercise helps to maintain quality of life, also inducing improvement of cognitive functions, stimulation of brain plasticity and resilience, in addition to promoting self-esteem and social interaction. The precise mechanisms by which exercise improves symptoms of depression are not fully clear, but it is probably multifactorial. In this project, the investigators aim to investigate variables that provide additional information about biomarkers involved in the pathophysiology of depression and therapeutic response to exercise. The investigators expect to find changes in biomarkers associated with potential mechanisms of neuroprotection (cytokines, markers of oxidative stress, Brain-derived neurotrophic factor (BDNF), cortisol) after exercise program and the role in the therapeutics of depression. To evaluate functional assessment indices will be used ergospirometry, a test that determines the respiratory, cardiovascular and metabolic activity. Overall, this project will help to investigate alternative adjunctive treatments for depression and their associated biomarkers with response.

ELIGIBILITY:
Inclusion Criteria:

* Major Depression Disorder According Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria
* Score higher or equal 18 in Hamilton Depression Rating Scale
* Age between 18 and 55 years old

Exclusion Criteria:

* Unstable Clinical Diseases
* Patients Unable to make Physical Exercises
* Present frequencies below 90% attendance in the program aerobic fitness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Physical exercise evaluation | One year
  Evaluate the physical exercise influence on the symptoms, according to HAM-D criteria, at the end of training program.

SECONDARY OUTCOMES:
Biomarkers level comparison | One year
  To compare possible levels of cytokines, before and after controled physical exercise.
Biomarkers level comparison | One year
  To compare possible levels of markers of oxidative stress, before and after controled physical exercise.
Biomarkers level comparison | One year
  To compare possible levels of BDNF (Brain-Derived Neurotrophic Factor), before and after controled physical exercise.
Biomarkers level comparison | One year
  To compare possible levels of Cortisol, before and after controled physical exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Machado-Vieira, Phd, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Siqueira CC, Valiengo LL, Carvalho AF, Santos-Silva PR, Missio G, de Sousa RT, Di Natale G, Gattaz WF, Moreno RA, Machado-Vieira R. Antidepressant Efficacy of Adjunctive Aerobic Activity and Associated Biomarkers in Major Depression: A 4-Week, Randomized, Single-Blind, Controlled Clinical Trial. PLoS One. 2016 May 6;11(5):e0154195. doi: 10.1371/journal.pone.0154195. eCollection 2016. PMID 27152523